CLINICAL TRIAL: NCT00308997
Title: Transcranial Magnetic Stimulation Guided by Neuroimaging for Patients With Persistent "Voices"
Brief Title: Transcranial Magnetic Stimulation for "Voices"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0409027023b; R01MH073673-01 (NIH); DATR A5-ETPD
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia; Hallucinations
Keywords: Auditory Hallucinations; Schizophrenia; Schizoaffective Disorder; Repetitive Transcranial Magnetic Stimulation; Wernicke's Area; Superior Temporal Gyrus
MeSH Terms: conditions — Schizophrenia; Hallucinations; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Active 1-hertz Repetitive Transcranial Magnetic Stimulation to Wernicke's area and right homologous area
  Interventions: Device: Active 1-Hertz Repetitive transcranial magnetic stimulation
- 2 (Sham Comparator): sham rTMS to Wernicke's area and a right homologous area
  Interventions: Device: 1-hertz Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: 1-hertz Repetitive Transcranial Magnetic Stimulation — Sham stimulation given to Wernicke's area or a right homologous area for 16 minutes per day x 5 days for week I, the same for week II with switch from right to left or left to right, and 5 more stimulation sessions (16 minutes per session) to the side producing greater benefit for week III.
  Other Names: Magstim Rapid-2
  Arms: 2
Device: Active 1-Hertz Repetitive transcranial magnetic stimulation — Active stimulation given to Wernicke's area or a right homologous area for 16 minutes per day x 5 days for week I, the same for week II with switch from right to left or left to right, and 5 more stimulation sessions (16 minutes per session) to the side producing greater benefit for week III.
  Other Names: Magstim Rapid-2
  Arms: 1

SUMMARY:
This study will determine the efficacy of MRI-guided transcranial magnetic stimulation (TMS)in reducing "voices" and other symptoms experienced by people with schizophrenia and schizoaffective disorder. In addition, the study will determine duration of improvement obtained during the course of trial participation via on-going monthly contact with study participants for up to 1 year after the trial.

DETAILED DESCRIPTION:
Schizophrenia is a severely disabling brain disorder that affects about 1% of the United States population. Approximately 50 to 80% of people with schizophrenia experience "voices," also known as auditory hallucinations. These hallucinations consist of spoken speech, which sometimes replicates the speaking voice of a familiar person, and sometimes reflects a speaking voice that is not known but becomes highly recognizable. The phrases and sentences expressed by "voices" are often highly disruptive, and may comment, cajole, criticize, and, in some cases, command the patient. They are often but not invariably distressing, and can disrupt one's ability to interact with others, work, study, and sleep. In about 25% of cases, medication treatment is either completely ineffective or only partially effective in relieving "voices." Effective treatment alternatives are needed to improve this troubling and often disabling symptom.

Recent studies have suggested that auditory hallucinations arise from parts of the brain that are ordinarily involved in perceiving actual spoken speech. Low frequency repetitive transcranial magnetic stimulation (rTMS), a technique that uses an electromagnet to induce reductions in cortical brain activity, may therefore be effective in quieting auditory hallucinations. The potential usefulness of this approach has been demonstrated by previous studies conducted at our medical center. This new study uses magnetic resonance imaging (MRI) to locate two areas of the brain involved in speech perception. These areas are in Wernicke's area in the left superior temporal gyrus, and in the right hemisphere in an analogous site in the superior temporal gyrus. Repetitive TMS is specifically positioned to reduce cortical excitability or reactivity at these two brain regions.

Participants in this double blind study will be randomly assigned to receive either real rTMS, or placebo stimulation, which feels similar to real rTMS but does not produce direct brain effects. Depending on group assignment, participation may last 4 to 8 weeks. Over the first 2 weeks, all participants will undergo two sequences of rTMS, each consisting of five 16-minute sessions. One sequence is directed to left Wernicke's area and the other sequence is directed to the right-sided equivalent area. During the third week, participants will receive five additional sessions to the left or right site that appeared to produce greater clinical improvement. All participants will then be informed as to whether they received real or placebo stimulation. Participants who received real stimulation will be offered 5 additional stimulation sessions at the brain site that achieved the best response. Participants who received placebo stimulation will be offered real stimulation for up to twenty sessions over 4 weeks using the same schedule described above. Assessments of severity of hallucinations and other clinical symptoms will be conducted after every fifth rTMS session by a clinician who does not know whether the participant is receiving real or placebo stimulation.

Neuropsychological testing will also be done before, during, and after the trial. Our previous trial demonstrated some improvement in verbal processing with no significant impairments in terms of memory, language or cognitive function. However, insofar as this trial involves a greater total "dose" of rTMS, careful monitoring of these functions is conducted throughout the trial.

In addition, the study will determine the degree to which improvement obtained during the course of trial is sustained over the ensuing months. This is accomplished via on-going monthly contact with study participants for up to 1 year after the last rTMS stimulation session.

ELIGIBILITY:
Inclusion Criteria:

* Auditory hallucinations that occur at least five times per day, on average
* Diagnosis of schizophrenia or schizoaffective disorder

Exclusion Criteria:

* Pregnant
* History of seizure that is not drug-induced or secondary to alcohol withdrawal
* Drug or alcohol abuse within 6 weeks of study entry (prior history of drug or alcohol abuse is not an exclusion)
* Changes in antipsychotic drug dosages within 4 weeks of study entry (patients do not need to be on antipsychotic medication to be included)
* Current significant untreated or unstable medical illness (e.g., poorly controlled diabetes mellitus, severe hypertension, unstable cardiac arrhythmia)
* Inability to understand the nature of the study due to severe psychotic disorganization, mental retardation, etc.
* Significant neurological condition (e.g., traumatic brain injury, multiple sclerosis)
* Factors that would preclude an MRI scan (e.g., severe obesity, claustrophobia, certain surgical implants with metallic components, metal shavings in the eye acquired while working as machinist)
* Cardiac pacemaker

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2006-02; Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph E. Hoffman, MD, Principal Investigator — Yale University School of Medicine, Department of Psychiatry
Locations (1):
- Yale Psychiatric Research, New Haven, Connecticut, United States

REFERENCES:
- [Background] Hoffman RE, Gueorguieva R, Hawkins KA, Varanko M, Boutros NN, Wu YT, Carroll K, Krystal JH. Temporoparietal transcranial magnetic stimulation for auditory hallucinations: safety, efficacy and moderators in a fifty patient sample. Biol Psychiatry. 2005 Jul 15;58(2):97-104. doi: 10.1016/j.biopsych.2005.03.041. PMID 15936729
- [Background] Hoffman RE, Boutros NN, Hu S, Berman RM, Krystal JH, Charney DS. Transcranial magnetic stimulation and auditory hallucinations in schizophrenia. Lancet. 2000 Mar 25;355(9209):1073-5. doi: 10.1016/S0140-6736(00)02043-2. PMID 10744097
- [Background] Hoffman RE, Cavus I. Slow transcranial magnetic stimulation, long-term depotentiation, and brain hyperexcitability disorders. Am J Psychiatry. 2002 Jul;159(7):1093-102. doi: 10.1176/appi.ajp.159.7.1093. PMID 12091184
- [Background] Poulet E, Brunelin J, Bediou B, Bation R, Forgeard L, Dalery J, d'Amato T, Saoud M. Slow transcranial magnetic stimulation can rapidly reduce resistant auditory hallucinations in schizophrenia. Biol Psychiatry. 2005 Jan 15;57(2):188-91. doi: 10.1016/j.biopsych.2004.10.007. PMID 15652879
- [Background] Chibbaro G, Daniele M, Alagona G, Di Pasquale C, Cannavo M, Rapisarda V, Bella R, Pennisi G. Repetitive transcranial magnetic stimulation in schizophrenic patients reporting auditory hallucinations. Neurosci Lett. 2005 Jul 22-29;383(1-2):54-7. doi: 10.1016/j.neulet.2005.03.052. Epub 2005 Apr 15. PMID 15936511
- [Background] Fitzgerald PB, Benitez J, Daskalakis JZ, Brown TL, Marston NA, de Castella A, Kulkarni J. A double-blind sham-controlled trial of repetitive transcranial magnetic stimulation in the treatment of refractory auditory hallucinations. J Clin Psychopharmacol. 2005 Aug;25(4):358-62. doi: 10.1097/01.jcp.0000168487.22140.7f. PMID 16012279
- [Background] Hoffman RE, Hampson M, Wu K, Anderson AW, Gore JC, Buchanan RJ, Constable RT, Hawkins KA, Sahay N, Krystal JH. Probing the pathophysiology of auditory/verbal hallucinations by combining functional magnetic resonance imaging and transcranial magnetic stimulation. Cereb Cortex. 2007 Nov;17(11):2733-43. doi: 10.1093/cercor/bhl183. Epub 2007 Feb 13. PMID 17298962
- [Derived] Hoffman RE, Wu K, Pittman B, Cahill JD, Hawkins KA, Fernandez T, Hannestad J. Transcranial magnetic stimulation of Wernicke's and Right homologous sites to curtail "voices": a randomized trial. Biol Psychiatry. 2013 May 15;73(10):1008-14. doi: 10.1016/j.biopsych.2013.01.016. Epub 2013 Feb 26. PMID 23485015
- See also: Click here for the Yale University website with information about this study — http://info.med.yale.edu/psych/clinics/rTMS.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Arm: Active 1-hertz Repetitive Transcranial Magnetic Stimulation to Wernicke's area and right homologous area
  Active 1-Hertz Repetitive transcranial magnetic stimulation : Active stimulation given to Wernicke's area or a right homologous area for 16 minutes per day x 5 days for week I, the same for week II with switch from right to left or left to right, and 5 more stimulation sessions (16 minutes per session) to the side producing greater benefit for week III.
- Placebo Arm: sham rTMS to Wernicke's area and a right homologous area
  1-hertz Repetitive Transcranial Magnetic Stimulation : Sham stimulation given to Wernicke's area or a right homologous area for 16 minutes per day x 5 days for week I, the same for week II with switch from right to left or left to right, and 5 more stimulation sessions (16 minutes per session) to the side producing greater benefit for week III.
Period: Overall Study
Arm/Group | Active Arm | Placebo Arm
Started | 56 | 29
Completed | 55 | 28
Not Completed | 1 | 1
Not completed — Subject feigned clinical data | 0 | 1
Not completed — Unable to tolerate intervention | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Arm | Placebo Arm | Total
Number analyzed (Participants) | 55 | 28 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (11.0) | 34.0 (10.0) | 35.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 15 | 44
  Male | 26 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Hallucination Change Score - Right (HCS-right)
Description: HCS score for participants assessed after 5 sessions, 16 minutes per session, who received either rTMS or sham stimulation delivered to the right superior temporal gyrus.
  HCS was anchored at 0 (corresponding to no AVHs), 10 (no change in hallucination severity) and 20 (AVHs twice as severe as baseline). Lower scores correspond to greater improvement
Time Frame: After 5 sessions of rTMS
Population: Subjects who did not complete the intervention were not analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 55 | 28
units on a scale | 7.78 (2.68) | 9.30 (1.47)

2. Primary Outcome: Hallucination Change Score - Left (HCS-left)
Description: HCS score for participants assessed after 5 sessions, 16 minutes per session, who received either rTMS or sham stimulation delivered to the left superior temporal gyrus.
  HCS was anchored at 0 (corresponding to no AVHs), 10 (no change in hallucination severity) and 20 (AVHs twice as severe as baseline). Lower scores correspond to greater improvement
Time Frame: After 5 sessions of rTMS
Population: Subjects who did not complete the intervention were not included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 55 | 28
units on a scale | 8.65 (2.74) | 8.50 (1.59)

3. Primary Outcome: Hallucination Change Score (HCS)
Description: HCS score assessed after 15 sessions, 16 minutes per session, delivered to both right superior temporal and left superior temporal gyrus sites using either rTMS or sham stimulation. For patients dropping out of the trial prematurely, last-observation-carried-forward data were used for this outcome variable.
  HCS was anchored at 0 (corresponding to no AVHs), 10 (no change in hallucination severity) and 20 (AVHs twice as severe as baseline). Lower scores correspond to greater improvement
Time Frame: After 15 sessions of rTMS
Population: Subjects who did not complete the intervention were excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 55 | 28
units on a scale | 6.45 (3.42) | 7.51 (2.26)

4. Secondary Outcome: Change in Hallucination Frequency
Description: AHRS frequency scale score assessed after 15 sessions, 16 minutes per session, of both right superior temporal and left superior temporal gyrus sites using either rTMS or sham stimulation (3 weeks). For patients dropping out of the trial prematurely, last-observation-carried-forward data were used for this outcome variable. The hallucination frequency range is from 0-9. The scores reported are difference scores, and an improvement is a higher score.
  Hallucination frequency is one of the variables incorporated into the AHRS (Auditory Hallucinations Rating Scale). The score is measured as change relative to baseline (i.e., baseline minus endpoint). Larger (positive) scores correspond to greater improvement.
Time Frame: After 15 sessions of rTMS
Population: Subjects who did not complete the intervention were excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 55 | 28
units on a scale | 1.31 (1.57) | 0.30 (1.61)

5. Secondary Outcome: Change in Total Auditory Hall Rating Scale (AHRS) Score
Description: Total AHRS score assessed after 15 sessions, 16 minutes per session, of both right superior temporal and left superior temporal gyrus sites using either rTMS or sham stimulation (3 weeks). For patients dropping out of the trial prematurely, last-observation-carried-forward data were used for this outcome variable. The score range is from 0-42. This is reported as a difference score and a higher score is an improvement.
  Total AHRS score is measured as change relative baseline (i.e., baseline minus endpoint). Larger (positive) scores correspond to greater improvement.
Time Frame: After 15 sessions of rTMS
Population: Subjects who did not complete the intervention were excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 55 | 28
units on a scale | 4.48 (6.90) | 3.0 (6.21)

6. Secondary Outcome: Clinical Global Improvement (CGI)Improvement
Description: CGI score assessed after 15 sessions, 16 minutes per session, of both right superior temporal and left superior temporal gyrus sites using either rTMS or sham stimulation (3 weeks). For patients dropping out of the trial prematurely, last-observation-carried-forward data were used for this outcome variable. The range for this score is from 1 to 7.
  Lower scores correspond to greater improvement
Time Frame: After 15 sessions of rTMS
Population: Subjects who did not complete the intervention were excluded from the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 55 | 28
units on a scale | 2.72 (1.15) | 3.21 (1.35)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the duration of the study, which was approximately 5 years.
Arm/Group | Active Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/28
Other Adverse Events (participants affected / at risk) | 30/55 | 5/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Arm (N=55) | Placebo Arm (N=28)
Somatic Discomfort (General disorders) | 14 | 4
Lightheaded/Dizziness (Nervous system disorders) | 5 | 0
Concentration Problems (Nervous system disorders) | 3 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Worsening Hallucinations/Audible Thoughts (Psychiatric disorders) | 5 | 1
Headache (Nervous system disorders) | 12 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes